CLINICAL TRIAL: NCT02216435
Title: Using Parkinson's Disease to Study the Role of the Substantia Nigra Pars Reticulata in Movement Initiation and Perception
Brief Title: Using Parkinson's Disease to Study the Role of the Substantia Nigra Pars Reticulata
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 13-2965; Univeristy of Colorado (Other Grant/Funding Number: 230 0894)
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Parkinson's Disease (PD) is a movement disorder causing either uncontrolled movement, slowness of movement, slowness of initiation of movement or rigidity of muscles. Deep Brain Stimulation (DBS) is the FDA-approved method for patients who no longer get effective treatment from the best available medication. The location in the brain where the electrode is placed during DBS surgery for PD is called the Subthalamic Nucleus or STN. This study aims to investigate another location in the brain, the Substantia nigra pars reticulata or SNr. The SNr is also known to be involved in motor control of muscles and may be involved in the process by which the initiation of movement occurs.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a movement disorder causing either uncontrolled movement, slowness of movement, slowness of initiation of movement or rigidity of muscles. One method of easing PD symptoms is the FDA-approved method of Deep Brain Stimulation (DBS) for patients who no longer get effective treatment from the best available medication. The location in the brain where the electrode is placed during DBS surgery for PD is called the Subthalamic Nucleus or STN. During placement of the DBS electrode, the patient is awake and is asked to do motor tasks to determine the correct placement in the STN and proper functioning of the DBS electrode. This study aims to investigate another location in the brain, the Substantia nigra pars reticulata or SNr, during the normal placement of the DBS electrode. This location is also known to be involved in motor control of muscles and may be involved in the process by which the initiation of movement occurs. The path through the brain to the STN used for DBS surgery goes into the SNr but currently, no testing of the SNr is performed. We will conduct a simple and well documented visual motor test to document the patient's stimulus perception and motor intention both at rest and during neural stimulation of the SNr.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease
* must be able to undergo awake surgery DBS
* must have unaided vision to view visual motor task

Exclusion Criteria:

* corrective eyeglasses or contact lenses

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease who are candidates for Deep Brain Stimulation surgery.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2014-07; Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

PRIMARY OUTCOMES:
Activity of the SNr | Immediately during Deep Brain Stimulation Surgery
  Recording and evaluating brain activity from the SNr (Substantia Nigra Pars Reticulata) in Parkinson's disease patients while the patient is undergoing the visual motor testing during Deep Brain Stimulation Surgery.

CONTACTS AND LOCATIONS:
Overall Officials: John A Thompson, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States